CLINICAL TRIAL: NCT02111902
Title: Determinants and Consequences of Low Vitamin D in Populations of African Descent
Brief Title: Vitamin D Ancillary Study in 5 Populations of African Origin
Acronym: VIDA
Status: Withdrawn | Type: Observational
Why Stopped: At the direction of our IRB, this project was incorporated into an existing study, LU#200038, NCT#02925156
Sponsor: Loyola University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Kwame Nkrumah University of Science and Technology (Other); University of Cape Town (Other); The University of The West Indies (Other); University Institute of Social and Preventive Medicine, Switzerland (Unknown); University of Washington (Other); Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Ramon Durazo, Professor, Loyola University
Other Study IDs: 202538; 1R01DK090360-01A1 (NIH)
Record Dates: First submitted 2014-04-04; First posted 2014-04-11 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Cardiovascular Disease; Obesity
Keywords: Cardiovascular Disease; Obesity; Physical Activity; Vitamin D deficiency; African Americans
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Motor Activity; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Serum Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The availability of data on plasma 25-Hydroxyvitamin D (25(OH)D) concentrations in the last two rounds of the National Health and Nutrition Examination Survey (NHANES) has generated a high level of interest in the consequences of 25(OH)D deficiency and in particular its potential impact on black Americans. Fundamental new questions about the biology of vitamin D have now come to the fore. Are low 25(OH)D-intact parathyroid hormone (iPTH) levels a physiologic "abnormality" in African Americans or does the 25(OH)D-iPTH system have sufficient plasticity to adapt to low sunlight exposure? Could the low 25(OH)D levels which result from the "gene- environment discordance" observed in dark skinned populations in the US be a risk factor for metabolic disorders? Ultimately, the public health community and regulatory bodies must offer recommendations for optimal levels and supplementation. The investigators propose to utilize cohorts from an ongoing NIH-funded study designed to identify determinants of weight change and cardiovascular disease risk in five Afro-origin populations [Modeling the Epidemiologic Transition Study (METS)] to examine these questions. The five METS countries include Ghana, Seychelles, South Africa, Jamaica and the US; the five populations differ greatly in terms of sun exposure and dietary intakes. In addition to the extensive energy expenditure, dietary intake and obesity-related metabolic markers being measured in METS, the investigators propose to assess plasma 25(OH)D, iPTH, serum and urinary calcium, plasma markers of bone resorption and formation, and quantitative ultrasound of the calcaneus. The associations of adiposity, weight change, cardiovascular disease (CVD) risk factors such as blood pressure and insulin, and bone strength with 25(OH)D and iPTH will be assessed. The proposed study will provide a comprehensive assessment of the distribution and determinants of 25(OH)D-iPTH and related physiologic measures across a wide range of latitude and lifestyles. These data should contribute substantially to the understanding of the "normal" range within which these hormones function and their significance in Afro- origin populations.

DETAILED DESCRIPTION:
Through its key role in bone mineral metabolism vitamin D deficiency was one of the first nutritional deficits linked to a clinical disease. A range of population and clinical research has now implicated less severe vitamin D deficiency as a potential risk factor for several chronic diseases [Melamed, et al. J Am Soc Nephrol 2009;20:2631-9; Michos et al. Future Cardiol, 2009;5:15-8; Reis et al. Diabetes Metab, 2005;31:318-25] and all-cause mortality [Melamed et al. Arch Intern Med, 2008;168:1629-37; Durazo-Arvizu et al. International Workshop on Statistical Modeling(IWSM);2010] is significantly increased at the low end of the 25(OH)D distribution among blacks and whites in the follow-up data from NHANES III. One out of 2 adults in the US has a 25(OH)D serum level < 30 ng/ml [Ginde et al. Arch Intern Med, 2009;169:626-32], currently considered the threshold for health-promoting levels [Howe et al. N Engl J Med, 2007;357:1981-2]. Light skin facilitates formation of 25(OH)D and consequently only 3% of US blacks have "optimal" levels, with very low levels (<10 ng/mL) found in 29% of blacks, compared to 5% of whites and10% of Mexican Americans [Ginde et al. Arch Intern Med, 2009;169:626-32]. Concern exists therefore that low serum levels of 25(OH)D may contribute to the disproportionately high risk for some chronic diseases in US blacks (eg, obesity, hypertension and CVD) [Pilz et al. Nat Rev Cardiol, 2009;6:621-30; Wang et al. Circulation, 2008;117:503-11]. At the present time the most convincing body of data on 25(OH)D and risk of chronic disease exists for obesity; the study proposed here will be conducted as an extension of a major international project on determinants of weight gain in Afro-origin populations.

25(OH)D has regulatory functions in several physiologic systems. Paradoxically, while US blacks have relatively lower serum 25(OH)D they have higher bone mineral density (BMD) and lower fracture rates, suggesting important variation in metabolic set points across populations [Aloia, Am J Clin Nutr, 2008;88:545S-550S]. However, it is not known if US blacks are at increased risk from the non-skeletal effects of low 25(OH)D. The overall health consequences of this shift in 25(OH)D levels and the threshold of "normal" for US blacks are thus unknown. The primary aim of this study is therefore to define the optimal level of 25(OH)D and the appropriate threshold for supplementation in the multi-ethnic US population. These data could have an important impact on public health recommendations regarding health-promoting levels of 25(OH)D.

Vitamin D levels in West Africans are similar to US whites, and much higher than in US blacks (see preliminary data). These cross-population contrasts represent one of the most significant known examples of a gene-environment interaction. By sampling Afro-origin populations across a range of latitudes, Ca++ intake, diet patterns, and lifestyles the investigators will model the determinants of 25(OH)D and related health effects. This research will incorporate 3 novel aspects. First, data on 25(OH)D will be standardized and a set of key determinants of 25(OH)D levels from 5 geographically separated populations of African descent will be available. Second, the study will generate precise covariate measures for obesity and other CV traits to test prospectively the association with 25(OH)D. Third, the investigators will have DXA measurements to examine 25(OH)D - PTH - bone density relationships and address a fundamental question about regulation of mineral metabolism and bone health. A major strength of this study will be state-of-the-art measurements of covariates for obesity, including doubly labeled water, activity monitoring, body composition and dietary intake. The role of 25(OH)D in obesity risk can therefore be evaluated with control for all of the key determinants of energy balance.

This study will utilize existing data and fasting samples from an ongoing NIH-funded study [Modeling the Epidemiologic Transition Study (METS; DK080763)]. METS began recruiting 2500 adults of African ancestry ages 25-45 from 5 countries (500 each from the US, Jamaica, Seychelles, South Africa, and Ghana) in October 2009. This study extends the follow-up period currently funded by METS to 6.2 years and uses a combined cohort-ecologic design to examine within-person and between-group associations.

Specific Aims:

1. Measure serum 25(OH)D and intact parathyroid hormone (iPTH) levels in 500 adults from the 5 METS sites (total N=2,500) at baseline and determine associations with latitude, diet, physical activity, adiposity, blood pressure (BP), and biochemical risk factors for CVD (eg, insulin, glucose, adiponectin, leptin, cholesterol).
2. Examine the association between baseline serum 25(OH)D and iPTH levels and changes in body composition and blood pressure over 6.2 years of follow-up.
3. Repeat measurement of serum 25(OH)D and iPTH at third follow-up examination (approximately 3.5 years after baseline) and measure BMD using DXA in the available cohort.

ELIGIBILITY:
Inclusion Criteria:

* Ages 25-44

Exclusion Criteria:

* Pregnant women will be excluded

Ages: 25 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A community-based probability sampling strategy is being used to recruit 500 adults, ages 25-44, from metropolitan Chicago, Spanish Town Jamaica, rural Ghana near Kumasi, Cape Town South Africa, and the Seychelles in the Indian Ocean
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-09 (Estimated); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
25-Hydroxyvitamin D | Baseline
Parathyroid Hormone (iPTH) | Baseline
Blood Pressure | Baseline, 2.5 years
Body Composition | Baseline, 2.5 years
  Body composition is estimated using bioelectrical impedance analysis (BIA) and race/sex specific equations. However, all participants will have body composition also measured using DXA (Dual energy x-ray absorptiometry).
Dietary Intake | Baseline, 2.5 years
  Each participant will complete at least two 24-hour recalls using the multiple pass method during each examination, one at the initial clinic visit and the second when the activity monitor is collected.
Physical Activity | Baseline, 2.5 years, 4 years
  Accelerometer
Bone Mineral Density | 2.5 years
  Dual energy x-ray absorptiometry (DXA) is a densitometry technique which provides a two-dimensional image of the bone being measured, to produce bone mineral density (BMD) values (mass of bone tissue per unit area).

SECONDARY OUTCOMES:
Serum Calcium | Baseline, 2.5 years
Serum Albumin | Baseline, 2.5 years
Urinary Calcium | Baseline, 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ramon A Durazo-Arvizu, PhD, Principal Investigator — Loyola University Chicago
Locations (5):
- Department of Public Health Sciences; Loyola University Chicago, Maywood, Illinois, United States
- Kwame Nkrumah University of Science and Technology, Kumasi, Ghana
- University of the West Indies, Kingston, Jamaica
- University Institute of Social and Preventive Medicine, Victoria, Seychelles
- University of Cape Town, Cape Town, South Africa

REFERENCES:
- [Derived] Durazo-Arvizu RA, Camacho P, Bovet P, Forrester T, Lambert EV, Plange-Rhule J, Hoofnagle AN, Aloia J, Tayo B, Dugas LR, Cooper RS, Luke A. 25-Hydroxyvitamin D in African-origin populations at varying latitudes challenges the construct of a physiologic norm. Am J Clin Nutr. 2014 Sep;100(3):908-14. doi: 10.3945/ajcn.113.066605. Epub 2014 Jul 9. PMID 25008852